CLINICAL TRIAL: NCT06822738
Title: A Prospective, Multicenter Clinical Study to Evaluate the Safety and Effectiveness of Gel Stent (XEN63) Implantation Using Ab Interno and Ab Externo Approaches in Subjects With Glaucoma
Brief Title: A Study to Assess Adverse Events and Effectiveness of Gel Stent (XEN63) Implantation Using Ab Interno and Ab Externo Approaches in Adult Participants With Glaucoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M22-087
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma; AGN-9003
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- XEN63 Ab Externo (Experimental): Participants will be implanted with XEN63 via ab externo surgical approach in the study eye. Participants will be followed for up to 12 months.
  Interventions: Device: XEN63 Glaucoma Treatment System
- XEN63 Ab Interno (Experimental): Participants will be implanted with XEN63 via ab interno surgical approach in the study eye. Participants will be followed for up to 12 months.
  Interventions: Device: XEN63 Glaucoma Treatment System

INTERVENTIONS:
Device: XEN63 Glaucoma Treatment System — Gel Stent

SUMMARY:
Glaucoma is the second most common cause of blindness in the world, second only to cataracts. This study will assess how safe and effective a glaucoma gel stent is when implanted using the ab interno (inside the eye) and ab externo (outside the eye) approach. Adverse events and intraocular pressure will be assessed.

XEN63 is an investigational device for the treatment of intraocular pressure (IOP) in patients with glaucoma when both medical and conventional surgical treatments have failed (for US approval) and when medical treatments have failed (for outside US [OUS] approval). Participants will be placed in one of two groups called study arms. One group will receive the XEN63 gel stent ab interno (inside the eye) and the other group will receive the XEN63 gel stent ab externo (outside the eye). Approximately 130 participants aged 45 years or older with glaucoma will be enrolled in this study at approximately 32 sites in the United States.

Participants will receive XEN63 implanted using either the ab interno approach or the ab externo approach on Day 1 and will be followed for 12 months.

Participants will attend regular visits during the study at a hospital or clinic. The safety and effect of the gel stent on your glaucoma will be checked by medical assessments and eye examinations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma in the study eye (SE) (meeting criterion a or b)

  1. That meets the following refractory glaucoma criteria of eyes diagnosed with glaucoma uncontrolled by maximal medical therapy (four or more classes of intraocular pressure (IOP)-lowering medications, or fewer in cases where it has been documented that certain medication classes cannot be tolerated or are contraindicated), and failed one or more incisional intraocular glaucoma surgeries (e.g., glaucoma filtering surgery, tube shunt)
  2. Uncontrolled by medical therapy (to meet out-of-US [OUS] requirements) with participants who only have glaucoma uncontrolled by medical therapy (non-refractory glaucoma), a maximum of 10 participants who meet only criterion b (and not a) will be enrolled in each cohort.

     Exclusion Criteria:
* History of angle-closure glaucoma where the angle has not been surgically opened in the SE.
* History of secondary open-angle glaucoma (e.g., neovascular, pigmentary, pseudoexfoliative, uveitic, angle recession/traumatic glaucoma, etc.) in the SE.
* Active inflammation (e.g., blepharitis, conjunctivitis, keratitis, uveitis) in the SE.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment Response of Achieving ≥ 20% Reduction in Intraocular Pressure (IOP) From Baseline on the Same or Fewer Number of IOP-Lowering Medications Compared to Baseline | Month 12
  IOP is a measurement of the fluid pressure inside the study eye. Treatment response is defined as IOP reduction on the same or fewer number of topical IOP-lowering medications.
Number of Participants with Adverse Events (AEs) | Month 12
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Mean Diurnal IOP | Month 12
  IOP is a measurement of the fluid pressure inside the eye. The mean diurnal IOP was the average of the IOP values of the study eye at Month 12.
Change From Baseline in Diurnal IOP | Baseline to Month 12
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Change from Baseline in Number of Topical IOP-Lowering Medications | Baseline to Month 12
  A numerical count by class of drug of topical IOP lowering medications being taken.
Mean Number of Topical IOP-Lowering Medications | Month 12
  A numerical count by class of drug of topical IOP lowering medications being taken.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (21):
  - Arizona Advanced Eye Research Institute /ID# 268363, Glendale, Arizona
  - LA Glaucoma Group /ID# 268444, Culver City, California
  - North Bay Eye Associates /ID# 277071, Petaluma, California
  - University Of Colorado - Anschutz Medical Campus /ID# 269947, Aurora, Colorado
  - Colorado Eye Institute /ID# 277072, Colorado Springs, Colorado
  - Brandon Eye Associates - Brandon /ID# 277074, Brandon, Florida
  - New Vision Eye Center /ID# 269955, Vero Beach, Florida
  - Coastal Research Associates - Roswell /ID# 268458, Roswell, Georgia
  - Illinois Eye Center - Peoria Location /ID# 277127, Peoria, Illinois
  - Stiles Eyecare Excellence & Glaucoma Institute /ID# 268451, Overland Park, Kansas
  - Minnesota Eye Consultants - Minneapolis /ID# 272445, Minneapolis, Minnesota
  - Vance Thompson Vision - Omaha /ID# 271599, Omaha, Nebraska
  - Oklahoma Eye Surgeons /ID# 269174, Oklahoma City, Oklahoma
  - Ophthalmic Partners of PA /ID# 276059, Bala-Cynwyd, Pennsylvania
  - Wills Eye Hospital Glaucoma Dept /ID# 268569, Philadelphia, Pennsylvania
  - Glaucoma Associates Of Texas /ID# 268745, Dallas, Texas
  - UT Southwestern Medical Center /ID# 268571, Dallas, Texas
  - El Paso Eye Surgeons /ID# 268356, El Paso, Texas
  - Berkeley Eye Center - Houston Greenway Plaza /ID# 277078, Houston, Texas
  - University of Virginia /ID# 277487, Charlottesville, Virginia
  - Vistar Eye Center - Roanoke - South Jefferson Street /ID# 276119, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-087